CLINICAL TRIAL: NCT02475434
Title: Post-Discharge Evaluation of Human Milk Cream Study Infants at 18 to 24 Month CGA: A Randomized Trial of the Use of Human Milk Cream to Decrease Length of Stay in Extremely Premature Infants
Brief Title: Use of Human Milk Cream to Decrease Length of Stay in Extremely Premature Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Prolacta Bioscience (Industry); Medical University Innsbruck (Other); The University of Texas Health Science Center, Houston (Other); Michigan State University (Other); Akron Children's Hospital (Other); Timpanogos Regional Hospital (Unknown); Orlando Health, Inc. (Other); St. Louis Children's Hospital (Other); Baylor Scott and White Health (Other); Westchester Medical Center (Other); Unity Health Toronto (Other); St. John Hospital & Medical Center (Other); Texas Tech University Health Sciences Center, El Paso (Other); Cook Children's Medical Center (Other); University of Oklahoma (Other)
Responsible Party: Principal Investigator, Amy Hair, Assistant Professor, Pediatrics-Neonatology, Director of Neonatal Nutrition, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-37231
Record Dates: First submitted 2015-06-05; First posted 2015-06-18 (Estimated); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: Human Milk; Prematurity; Nutrition; Human Milk Cream
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cream Supplement group (Experimental): Infants randomized to the cream supplement group will receive an exclusive HM-based diet with the addition of a HM-derived cream caloric supplement.
  Interventions: Dietary Supplement: Cream Supplement group
- Control Group (No Intervention): Infants randomized to the Control group will receive the standard regimen of an exclusive HM-based diet (no cream supplement).

INTERVENTIONS:
Dietary Supplement: Cream Supplement group — Infants in the intervention arm will receive the cream supplement in addition to the standard regimen.
  Other Names: ProlactCR
  Arms: Cream Supplement group

SUMMARY:
At present, widespread use of the human milk-based caloric supplement (cream) has not occurred, particularly in infants with bronchopulmonary dysplasia (BPD), and further data are needed to support its adoption as a standard care practice.

The investigators hypothesize that infants who receive an exclusive human milk (HM)-based diet with the addition of a HM-derived cream caloric supplement (Cream group) will have a shorter length of initial hospital stay compared to infants receiving the standard regimen of an exclusive HM-based diet (Control group). The investigators hypothesize that the effects of the cream caloric supplement will be greater in the subgroup of infants who develop BPD so the relationship will be evaluated between Cream Supplement study group and postmenstrual age (PMA) at discharge and the incidence of BPD. Investigators will also evaluate the post-hospital discharge growth, body composition, and neurodevelopmental outcomes at 18 to 24 months CGA of the infants 500-1250 grams BW who received an exclusive human milk diet including cream supplement or control in the NICU.

DETAILED DESCRIPTION:
The primary hypothesis of the study is that infants who receive an exclusive HM-based diet with the addition of a HM-derived cream caloric (Cream group) will have a shorter length of initial hospital stay compared to infants receiving the standard regimen of an exclusive HM-based diet (Control group).

The study design is a randomized controlled trial in preterm infants (birth weight 500-1250g) comparing the use of a human milk cream supplement added to an exclusive HM-based diet (Cream group) to an exclusive HM-based diet without the use of a cream supplement (Control group). Each study group will use mother's own milk, donor HM if needed (donor HM should be obtained from a Human Milk Banking Association of North America (HMBANA) or Prolacta milk bank that uses Holder method pasteurization and does not homogenize the milk) and a donor human milk-derived fortifier (Prolact+ H2MF®) according to the study feeding protocol. Feeding will be done by protocol in which fortification will begin when the baby is receiving 60 mL/kg/day of enteral nutrition. The randomization will be performed in blocks (block size to remain blinded) without the use of stratification variables except for study site. While blinding of study groups is always desirable in randomized studies, because of the nature of the interventions and the varying methods by which the nutrition is prepared and delivered in different units, this will not be possible for this study.

Sample Size:

The number of infants to be included in this study is based on the primary endpoint of a reduction in the length of hospital stay in days by 12.1 days with a standard deviation of 31 days. With a two-tailed 5% significance level and 80% power, a sample size of 210 (n=105 per group) is needed to demonstrate a difference of this magnitude between the 2 study groups.

Study Duration:

All study infants will be followed until discharge or transfer from the medical institution or death (hospital stay is an expected average of 10 weeks). Infants will be transitioned completely off an exclusive HM-based diet no earlier than 34 weeks PMA, however, infants will be followed until hospital discharge (total of an estimated average of 10 weeks) to collect anthropometric and study outcome data.

Study Population:

Each study subject must meet all of the indicated inclusion criteria and none of the exclusion criteria.

Study Procedure:

After eligibility of the infant is determined and informed consent is obtained from the parent or legal guardian, infants will be randomized using a stratified (by study site) block scheme noted above into either the group that will receive human milk cream (Cream Supplement) or not (Control). All study infants will follow the study feeding protocol. The use of fortifier, both the timing of initiation and advancing of feeds will be per study protocol as tolerated. Study infants are to receive only an exclusive HM-based diet and they are not to deviate from the protocol (receiving formula, medium chain triglyceride (MCT) oil, liquid protein supplement, bovine fortifier, etc). Once breast milk (either mother's or donor) fortification is initiated and infants reach feeds of at least 100 mL/kg/day, for infants randomized to the cream group, they will start receiving the cream supplement per protocol. HM cream supplement will be added to feeds to provide an additional 2 kcal/oz of energy (amount of cream to add equals amount of unfortified milk x 0.04 rounded to the nearest full mL). For example, 4 mL of cream would be added to 96 mL of unfortified milk and then the fortifier is added to the milk-cream mixture. The Control group will not receive cream and will be fed per Table 1. Infants will be followed and studied until discharge, transfer to a non-study institution, removal from the study or death. Starting no sooner than 34 weeks PMA, infants will be transitioned over 5 days to either mother's milk with bovine fortifier or transitional formula according to investigative site's standard of care. All infants will have a brain MRI at "term equivalent" age (if this is routine practice at the study site). Infants will also have body composition determined by dual energy x-ray absorptiometry (DXA) scan (if available at the study site). One outpatient study visit will occur at 18 to 24 months post discharge to obtain anthropometric data, interim medical history, demographic and socioeconomic information, and nutrition history of the child since discharge (formula, human milk, vitamins, and medications). A neurodevelopmental evaluation (The Bayley Scales of Infant Development III) will also be performed by a certified tester during this visit. In addition, data from NICU hospitalizations will be collected during this visit. Data collection will include: demographics (gestational age, birth weight, gender, and race), APGAR scores, nutrition and feeding related issues (parental nutrition and constituents, feeding regimen, feeding intolerance), growth parameters (weight, length, and head circumference), medications (caffeine, furosemide, chlorothiazide, hydrocortisone, dexamethasone, insulin, and dopamine), nutrition related labs, and morbidities (intraventricular hemorrhage, patent ductus arteriosus, necrotizing enterocolitis, spontaneous intestinal perforation, episodes of sepsis, chronic lung disease).

Anthropometric Measurements:

At each study site, designated study personnel (preferably no more than 3 consistent trained personnel), will be responsible for weekly anthropometric measurements. The personnel will be trained or will demonstrate proficiency in obtaining anthropometric measurements using proper equipment. They will take weekly weights, lengths using only a study length board to be provided, and head circumference measurements. Each measurement will be taken twice and the average of the two will be recorded (for the weekly measurement).

Human Milk Samples:

Three times a week (on 3 separate days), samples of the human milk (either mother's own or donor) per study infant will be obtained (4 mL in a syringe) and will be stored for future macronutrient analysis after study completion. The samples should be stored at -20 degrees C. The sample should be from a batch of unfortified human milk and should represent the milk to be used to prepare 24 hours of feedings. Stored samples will be sent to the coordinating study center for post-study analysis.

Microbiome Samples:

For all enrolled infants, tracheal aspirates (if intubated in the first 24 hours of life) and stool for post-study evaluation of infants' airway and gastrointestinal microbiome will be collected as feasible. A recent study by Lohmann et al showed that reduced diversity of the microbiome may be an important factor in the development of BPD. In addition, studies have shown that human milk positively affects the microbiome of premature infants. Tracheal aspirates will be obtained per study protocol if infants are intubated at birth to 24 hours of age, 48-72 hours of age, 7 days of age, and 28 days of age or at time of extubation if sooner. Any tracheal aspirate obtained within this time frame is acceptable (samples are of convenience with routine suctioning and care). Stool samples will be obtained per study protocol at the 1st, 2nd, 3rd, and 4th weeks of life. The infants' first stool (meconium) should be obtained. Samples will be collected and frozen at -80 degrees C and will be sent to the coordinating study center for post-study microbiome analysis.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight 500-1250g.
* Must be likely to be able to adhere to a feeding protocol involving mother's own milk/donor milk that will include fortification using HM-based product (Prolact+H2MF®) and, potentially, human milk-based cream supplement.
* Enteral feeding must begin before day 14 of life and parenteral nutrition must be started by day 2 of life.
* Informed consent obtained from parent or legal guardian prior to reaching 100 ml/kg/day of fortified feeds. Consent should be obtained as soon as possible for eligible infants to collect tracheal aspirates (if intubated) and meconium stool. However, consent must be obtained prior to reaching 100 ml/kg/day of fortified feeds because this is when randomization will occur.

Exclusion Criteria:

* Unlikely to survive the study period.
* Enrolled in another clinical study affecting nutritional management during the study period.
* Decision to not start minimum enteral feed before day 14 of life or parenteral nutrition before day 2 of life.
* Presence of clinically significant congenital heart disease or other major congenital malformation.
* Presence prior to enrollment of intestinal perforation or Stage 2 Necrotizing enterocolitis prior to tolerating fortified feeds.
* Reasonable likelihood of early transfer to a non-study institution.
* Unable to participate for any reason based on the decision of the study investigator.

Max Age: 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 210 (Actual)
Dates: Start 2015-06-10 (Actual); Primary Completion 2019-06-25 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
Length of Stay | From birth to death or discharge from the Neonatal ICU, assessed up to 5 months
  The primary endpoint for the study is the difference in length of hospital stay (days) between the two groups from birth until discharge or removal from the study (due to transfer to non-study institution or death), whichever comes first.

SECONDARY OUTCOMES:
Incidence of Bronchopulmonary dysplasia and relationship to postmenstrual age at discharge in infants who received cream supplement | From birth to death or discharge from the Neonatal ICU, assessed up to 5 months
  The secondary endpoint is to evaluate if Infants who have BPD and receive the cream supplement will be discharged home at an earlier postmenstrual age compared to infants with BPD who do not receive the cream supplement.

CONTACTS AND LOCATIONS:
Overall Officials: Amy B Hair, MD, Principal Investigator — Texas Children's Hospital, Baylor College of Medicine
Locations (8):
- United States (7):
  - Orlando Health, Inc. - Winnie Palmer Hospital for Women and Babies, Orlando, Florida
  - Michigan State University, East Lansing, Michigan
  - Children's Hospital Medical Center of Akron, Boardman, Ohio
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine / Texas Children's Hospital, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Wasatch Neonatal, Orem, Utah
- University Hospital, Innsbruck, Austria

REFERENCES:
- [Background] Schanler RJ. Outcomes of human milk-fed premature infants. Semin Perinatol. 2011 Feb;35(1):29-33. doi: 10.1053/j.semperi.2010.10.005. PMID 21255704
- [Background] Sullivan S, Schanler RJ, Kim JH, Patel AL, Trawoger R, Kiechl-Kohlendorfer U, Chan GM, Blanco CL, Abrams S, Cotten CM, Laroia N, Ehrenkranz RA, Dudell G, Cristofalo EA, Meier P, Lee ML, Rechtman DJ, Lucas A. An exclusively human milk-based diet is associated with a lower rate of necrotizing enterocolitis than a diet of human milk and bovine milk-based products. J Pediatr. 2010 Apr;156(4):562-7.e1. doi: 10.1016/j.jpeds.2009.10.040. Epub 2009 Dec 29. PMID 20036378
- [Background] Cristofalo EA, Schanler RJ, Blanco CL, Sullivan S, Trawoeger R, Kiechl-Kohlendorfer U, Dudell G, Rechtman DJ, Lee ML, Lucas A, Abrams S. Randomized trial of exclusive human milk versus preterm formula diets in extremely premature infants. J Pediatr. 2013 Dec;163(6):1592-1595.e1. doi: 10.1016/j.jpeds.2013.07.011. Epub 2013 Aug 20. PMID 23968744
- [Background] Abrams SA, Schanler RJ, Lee ML, Rechtman DJ. Greater mortality and morbidity in extremely preterm infants fed a diet containing cow milk protein products. Breastfeed Med. 2014 Jul-Aug;9(6):281-5. doi: 10.1089/bfm.2014.0024. Epub 2014 May 27. PMID 24867268
- [Background] Section on Breastfeeding. Breastfeeding and the use of human milk. Pediatrics. 2012 Mar;129(3):e827-41. doi: 10.1542/peds.2011-3552. Epub 2012 Feb 27. PMID 22371471
- [Background] Biniwale MA, Ehrenkranz RA. The role of nutrition in the prevention and management of bronchopulmonary dysplasia. Semin Perinatol. 2006 Aug;30(4):200-8. doi: 10.1053/j.semperi.2006.05.007. PMID 16860160
- [Background] Theile AR, Radmacher PG, Anschutz TW, Davis DW, Adamkin DH. Nutritional strategies and growth in extremely low birth weight infants with bronchopulmonary dysplasia over the past 10 years. J Perinatol. 2012 Feb;32(2):117-22. doi: 10.1038/jp.2011.67. Epub 2011 May 26. PMID 21617642
- [Background] Wojcik KY, Rechtman DJ, Lee ML, Montoya A, Medo ET. Macronutrient analysis of a nationwide sample of donor breast milk. J Am Diet Assoc. 2009 Jan;109(1):137-40. doi: 10.1016/j.jada.2008.10.008. PMID 19103335
- [Background] Vieira AA, Soares FV, Pimenta HP, Abranches AD, Moreira ME. Analysis of the influence of pasteurization, freezing/thawing, and offer processes on human milk's macronutrient concentrations. Early Hum Dev. 2011 Aug;87(8):577-80. doi: 10.1016/j.earlhumdev.2011.04.016. Epub 2011 May 17. PMID 21592688
- [Background] Hair AB, Blanco CL, Moreira AG, Hawthorne KM, Lee ML, Rechtman DJ, Abrams SA. Randomized trial of human milk cream as a supplement to standard fortification of an exclusive human milk-based diet in infants 750-1250 g birth weight. J Pediatr. 2014 Nov;165(5):915-20. doi: 10.1016/j.jpeds.2014.07.005. Epub 2014 Aug 15. PMID 25130571
- [Background] Walsh MC, Kliegman RM. Necrotizing enterocolitis: treatment based on staging criteria. Pediatr Clin North Am. 1986 Feb;33(1):179-201. doi: 10.1016/s0031-3955(16)34975-6. PMID 3081865
- [Background] Lohmann P, Luna RA, Hollister EB, Devaraj S, Mistretta TA, Welty SE, Versalovic J. The airway microbiome of intubated premature infants: characteristics and changes that predict the development of bronchopulmonary dysplasia. Pediatr Res. 2014 Sep;76(3):294-301. doi: 10.1038/pr.2014.85. Epub 2014 Jun 18. PMID 24941215
- [Background] Olsen IE, Groveman SA, Lawson ML, Clark RH, Zemel BS. New intrauterine growth curves based on United States data. Pediatrics. 2010 Feb;125(2):e214-24. doi: 10.1542/peds.2009-0913. Epub 2010 Jan 25. PMID 20100760
- See also: Product Description — https://www.prolacta.com/en/